CLINICAL TRIAL: NCT07186049
Title: Impact of Exercise Associated With Cognitive-behavioral Therapy in Smokers: a Randomized Clinical Trial
Brief Title: Impact of Exercise Associated With Cognitive-behavioral Therapy in Smokers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agnaldo José Lopes (Other)
Responsible Party: Sponsor-Investigator, Agnaldo José Lopes, Doctor with a PhD, Centro Universitário Augusto Motta
Organization: Centro Universitário Augusto Motta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 02565743750
Record Dates: First submitted 2025-09-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Smoking (Tobacco) Addiction
Keywords: Smoking; Physical exercise; Cognitive-behavioral therapy
MeSH Terms: conditions — Smoking; Behavior, Addictive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 3 General Health Guidelines. (Active Comparator): General Health Guidelines
  Interventions: Behavioral: General Health Guidelines
- Group 1 Thesis (Active Comparator): Thesis Sessions
  Interventions: Behavioral: Thesis Sessions
- Group 2 Thesis and Exercises (Active Comparator): Thesis Sessions + Home Exercises
  Interventions: Behavioral: Thesis and Exercises

INTERVENTIONS:
Behavioral: Thesis Sessions — Thesis Sessions
  Arms: Group 1 Thesis
Behavioral: General Health Guidelines — General Health Guidelines
  Arms: Group 3 General Health Guidelines.
Behavioral: Thesis and Exercises — Thesis and Exercises
  Arms: Group 2 Thesis and Exercises

SUMMARY:
Smoking remains one of the leading causes of global morbidity and mortality, responsible for more than 8 million deaths annually, according to data from the World Health Organization. In addition to its physical effects, such as cancer, cardiovascular, and respiratory diseases, tobacco use also negatively impacts mental health and quality of life (QoL). Despite public health measures, its prevalence remains high, especially among vulnerable groups, requiring integrated approaches that address both the physiological and psychological aspects of addiction.

This study aims to evaluate the effects of combining physical exercise and cognitive behavioral therapy (CBT) on smoking cessation. Specifically, it seeks to assess the effectiveness of a structured exercise program in promoting abstinence, improving physical and mental health, and reducing cigarette consumption, as well as analyzing the impacts on fatigue, lung function, exercise capacity, and quality of life of participants over a 12-week intervention.

Methodologically, a randomized clinical trial will be conducted with 66 smokers recruited from the Piquet Carneiro Polyclinic of the Rio de Janeiro State University. Participants will be randomly assigned to three groups: CBT alone, CBT combined with structured exercises, and a control group with general health counseling. Assessments will include spirometry, impulse oscillometry, the FACIT-Fatigue scale, the Fagerström test, a cardiopulmonary exercise test, and the SF-36 questionnaire, administered at three time points: baseline, 6 weeks, and 12 weeks.

The combination of exercise and CBT is expected to significantly increase abstinence rates, promoting improvements in physical and mental health parameters, reduced cigarette consumption, increased exercise capacity, improved lung function, and decreased fatigue. Furthermore, a reduction in anxiety and depression levels is expected, reflecting the effectiveness of behavioral strategies in modulating the psychological factors associated with smoking.

This study is highly relevant to Rehabilitation Sciences, as it proposes an integrated intervention that can support the development of more effective and holistic public health programs aligned with national targets and the Sustainable Development Goals. By exploring the interface between physical activity, mental health, and smoking cessation, it contributes to the training of more qualified health professionals and the advancement of patient-centered rehabilitation strategies, promoting sustainable benefits to public health.

DETAILED DESCRIPTION:
Detailed Description of the Thesis Title: Impact of Exercise Combined with Cognitive-Behavioral Therapy in Smokers: A Randomized Clinical Trial

Objectives

General Objective:

To evaluate the effects of combining physical exercise interventions with cognitive-behavioral therapy on smoking cessation among adult smokers.

Specific Objectives:

To assess the efficacy of a structured physical exercise program in promoting smoking cessation and improving the physical and mental health of participants.

To evaluate changes in smoking behaviors, including frequency and quantity of cigarettes smoked, during the clinical trial.

To analyze the effects of the combined intervention on general fatigue, lung function, and exercise capacity.

To measure the quality of life (QoL) of smokers before and after the intervention, considering physical, emotional, and social aspects.

Scientific Rationale and Relevance The scientific relevance of this study lies in its potential to inform the development of integrated rehabilitation strategies that address both cessation and the sequelae of tobacco use. The research aligns with national health priorities, particularly those related to chronic non-communicable diseases (NCDs), and supports the Sustainable Development Goals (SDGs) of the United Nations, notably SDG 3 (Good Health and Well-being). By focusing on the intersection of physical activity, mental health, and tobacco cessation, the study aims to contribute to the formation of better-trained health professionals and the development of patient-centered, holistic public health policies.

Methodology Study Design This is a randomized, controlled, parallel-group clinical trial with a 12-week intervention period. The study will be conducted at the Piquet Carneiro University Polyclinic (PPC), State University of Rio de Janeiro (UERJ), Brazil. The protocol will be preregistered on ClinicalTrials.gov to ensure methodological transparency and reproducibility.

Sample and Recruitment A total of 66 adult smokers will be recruited from the Anti-Smoking Program Outpatient Clinic at PPC-UERJ. The inclusion criteria are: age 18 years or older, clinical diagnosis of active smoking (combustible cigarettes), and availability to participate in all phases of the study. Exclusion criteria include unstable cardiac conditions, severe orthopedic problems, cognitive disorders that may interfere with participation, and concurrent involvement in other cessation or behavioral intervention studies.

Recruitment will be systematic, with the collaboration of the clinic's medical staff to ensure a diverse and representative sample. The sample size was calculated using G*Power 3.1, considering a one-way ANOVA with three independent groups, a significance level of 0.05, statistical power of 80%, and a large effect size (f = 0.40). To account for potential dropouts (estimated at 20%), the final sample size may be increased to approximately 81 participants.

Randomization and Groups

Participants will be randomly allocated into three parallel groups using block randomization with a specific software tool:

Group 1 (CBT): Participants receive only cognitive-behavioral therapy, focusing on behavioral modification strategies and motivational interviewing.

Group 2 (CBT + Exercise): Participants receive both CBT and a structured, supervised physical exercise program, including home-based sessions and weekly remote follow-up.

Group 3 (Control): Participants receive only general health education, with no supervised exercise or CBT.

Interventions CBT Protocol: Weekly sessions, based on motivational interviewing and the Stages of Change Model (Prochaska and DiClemente), addressing the psychological and behavioral aspects of tobacco dependence. The intervention is tailored to the individual's readiness to change, focusing on goal setting, overcoming barriers, and reinforcing positive behaviors.

Exercise Protocol: Home-based functional and aerobic exercise sessions, three times per week for 12 weeks, including warm-up, muscle strengthening, postural control, aerobic circuits, and stretching. Adherence is monitored via activity logs and weekly video submissions.

Control Group: Receives standard health advice only. Assessments Assessments are conducted at three time points: baseline (week 0), intermediate (week 6), and post-intervention (week 12). All instruments used are validated for the target population and administered by trained staff.

Clinical Evaluation: Sociodemographic data, medical history, smoking habits, and physical examination.

Fatigue Assessment: FACIT-Fatigue Scale (FACIT-F), a 13-item Likert scale measuring perceived fatigue.

Quality of Life: SF-36 questionnaire, covering physical, emotional, and social domains.

Pulmonary Function: Spirometry (measuring FVC, FEV1, FEV1/FVC, FEF25-75%) and impulse oscillometry (measuring respiratory resistance and reactance at various frequencies).

Nicotine Dependence: Fagerström Test for Nicotine Dependence (FTND), a 6-item scale.

Exercise Capacity: Cardiopulmonary exercise testing (CPET) using FitMate™ PRO, measuring peak oxygen consumption (VO2peak), ventilatory parameters, and functional reserve.

Adherence and Safety: Monitored throughout the study, with protocols for managing adverse events and withdrawal criteria.

Outcomes

Primary Outcome:

Smoking cessation rate, defined as the percentage of participants who remain abstinent during the follow-up period, confirmed by self-report and biochemical verification (cotinine levels and/or exhaled CO).

Secondary Outcomes:

Reduction in frequency and quantity of cigarettes smoked. Improvements in exercise capacity (VO2peak), pulmonary function, and general fatigue.

Enhanced quality of life (SF-36 scores). Changes in nicotine dependence (FTND scores). Adherence to intervention protocols. Data Analysis

Data will be managed in Microsoft Excel® and analyzed using IBM SPSS Statistics® (version 26.0). Statistical analyses include:

Descriptive statistics for all variables. Normality testing (Shapiro-Wilk). ANOVA for group comparisons (parametric data), Kruskal-Wallis for non-parametric data.

Chi-square or Fisher's exact test for categorical data. Post-hoc analyses (Tukey or Dunn with Bonferroni correction) for significant group differences.

Repeated measures ANOVA or Friedman test for within-group comparisons over time.

Logistic regression for analyzing the association between intervention type and smoking cessation, adjusting for covariates.

ANCOVA for secondary outcomes, controlling for baseline values. Significance set at p < 0.05, with 95% confidence intervals. Ethical Considerations The research protocol will be submitted to the Ethics Committee via Plataforma Brasil, in compliance with Resolution 466/2012 of the National Health Council and Law No. 14.874/2024 on human research. All participants will provide informed consent and will be assured of confidentiality, the right to withdraw, and access to clinical or psychological care if needed. The study includes provisions for reimbursement of travel expenses in cases of financial hardship and protocols for managing unexpected risks or adverse events.

Funding and Timeline The study is funded by the Brazilian Coordination for the Improvement of Higher Education Personnel (CAPES). The timeline includes project development, ethical approval, data collection, analysis, manuscript preparation, and dissemination of results over a period from 2025 to 2028.

Expected Results It is anticipated that the combined intervention group (CBT + Exercise) will demonstrate a significantly higher smoking abstinence rate compared to the control group, along with greater improvements in physical capacity, pulmonary function, fatigue reduction, and quality of life. The study also expects to observe positive changes in mental health parameters, such as reduced anxiety and depression, and increased adherence to healthy behaviors.

The findings will provide evidence to support the integration of physical and behavioral interventions in tobacco cessation programs, potentially influencing clinical practice guidelines and public health policy. The research aims to bridge gaps in current knowledge regarding the synergistic effects of exercise and CBT, contributing to more effective, patient-centered rehabilitation strategies.

Hypothesis:

This doctoral research presents a rigorous, innovative approach to smoking cessation, integrating physical exercise and cognitive-behavioral therapy within a randomized clinical trial framework. By addressing both the physiological and psychological dimensions of tobacco dependence, the study seeks to generate robust evidence to inform the design of holistic, sustainable health interventions. The expected outcomes have the potential to reduce the burden of smoking-related diseases, improve individual and population health, and support the development of more effective public health policies.

ELIGIBILITY:
Inclusion criteria:

* Participants 18 years of age or older;
* Clinical diagnosis of active smoking of combustible cigarettes;

Exclusion criteria:

* Unstable heart disease or severe orthopedic problems;
* Cognitive disorders that may interfere with understanding and participation in behavioral interventions;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-10-22 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The smoking cessation rate | 12 weeks
  The primary outcome of this study is the smoking cessation rate, defined as the percentage of participants who remain abstinent from tobacco use during the follow-up period. To ensure the robustness of the results, abstinence will be verified by participants' self-reports and confirmed by biochemical measures performed by physicians, such as blood cotinine levels and/or exhaled carbon monoxide (CO) testing. The selection of this primary outcome is based on the clinical relevance of achieving smoking cessation, as it contributes to improved individual health and serves as a direct indicator of the effectiveness of the proposed combined intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Agnaldo J José, Principal Investigator — Augusto Motta University Center
Locations (1):
- PPC/UERJ - Piquet Carneiro University Polyclinic, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
I'm still not sure; I will talk to my advisor